CLINICAL TRIAL: NCT01723293
Title: Effect of a Specific Exercise Program During Whole Pregnancy on Fetal Heart Rate Response to Maternal Effort in Third Trimester. A Randomised Controlled Trial
Brief Title: Fetal Cardiovascular Response to Maternal Exercise During Third Trimester
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, María Perales Santaella, PhD Student, Technical University of Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Fetal responses to exercise
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2012-08

CONDITIONS: Pregnancy
Keywords: Fetal heart rate, pregnancy, fetus, cardiovascular system

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Sedentary pregnant women
- Exercise group (Experimental)
  Interventions: Behavioral: Exercise group

INTERVENTIONS:
Behavioral: Exercise group — The physical conditioning program included a total of three 55-60 minute sessions per week. Pregnant women started in 9-12 weeks and finished in 38-40 weeks, therefore, an average of 85 training sessions were planned for each participant. All subjects wore a heart rate (HR) monitor (Polar FT7, Finland) during the training sessions to ensure that the exercise intensity was light to moderate.
  Each session included a 25-minutes of aerobic exercise, 10-minutes of strength exercise and balance exercise as well, and 10-minutes of pelvic floor muscles training.
  Arms: Exercise group

SUMMARY:
The purpose of this study was to examine the behavior of the fetal heart rate in response to different intensities of acute maternal exercise in training and non-training pregnant women

DETAILED DESCRIPTION:
Fetal heart rate is considered an important index of fetal well-being, especially during the third trimester of pregnancy (Rodney JR, Huntley BJ, Rodney WM, 2012). An increase in the FHR of 5-25 beats per min (bpm) in response to maternal exercise has been established as a normal reaction(Riemann,Kanstrup Hansen, 2000)however the normal FHR response to maternal exercise has remained unclear for several reasons

Most of the studies are focused on obtain data in order to examine the fetal heart rate response to maternal exercise using cardiotocography measurements prior to and following maternal exercise

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines
* Being able to communicate in spanish
* Giving birth at Hospital Universitario de Fuenlabrada

Exclusion Criteria:

* Multiparity
* Obstetrician complications
* Being interested in the study after 18 weeks
* Not being regular in physical exercise program
* Younger than 18 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-05 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Fetal heart rate | Up to 34 weeks
  Fetal heart rate was measured before and after maternal walking exercise at 40 and 60% MaxHR

SECONDARY OUTCOMES:
Fetal outcomes | After labor
  Birth weight
Maternal outcomes | During labor
  Type of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Barakat, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politecnica de Madrid, Madrid, Madrid, Spain